CLINICAL TRIAL: NCT05556850
Title: Efficacy of STABL Virtual Rehabilitation: A Randomized Controlled Study
Brief Title: Efficacy of STABL Virtual Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-00951
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Physical Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation using STABL platform (Experimental): Patients undergoing minor knee procedures (defined as meniscectomy and synovectomy) will be randomized to virtual rehabilitation using the STABL platform
  Interventions: Behavioral: STABL Virtual Rehabilitation
- Rehabilitation using standard physical therapy (No Intervention): Patients undergoing minor knee procedures (defined as meniscectomy and synovectomy) will be randomized to standard physical therapy.

INTERVENTIONS:
Behavioral: STABL Virtual Rehabilitation — STABL is a digital health platform that uses computer-vision technology to facilitate at-home post-op recovery for patients while enabling remote monitoring by their surgeon. The platform is fully HIPAA compliant.
  STABL analyzes a patient's biomechanics in real time while they perform their recovery exercises to provide them with cues to ensure the exercises are done correctly and track adherence. They then relay all the data to the patient's clinician to allow them to monitor their recovery remotely, address any adherence barriers, and mitigate readmission risks that arise in a more timely manner.
  Arms: Rehabilitation using STABL platform

SUMMARY:
The purpose of the proposed study is to evaluate the efficacy of STABL rehabilitation vs in-person rehabilitation following meniscectomy or synovectomy. STABL is a digital health platform that uses computer-vision technology to facilitate at-home post-op recovery for patients while enabling remote monitoring by their surgeon.

DETAILED DESCRIPTION:
Patients undergoing minor knee procedures (defined as meniscectomy and synovectomy) will be randomized to virtual rehabilitation using the STABL platform or standard physical therapy over the course of 6 weeks to determine any possible difference in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Underwent meniscectomy or synovectomy surgery
* Age 18-65
* Ability to comply with a standardized postoperative protocol
* Willing and able to provide consent

Exclusion Criteria:

* Previous knee surgery
* Patients at any increased risk of falls or at increased risk from harm due to falling, including issues with vertigo, osteoporosis, or a history of past falls
* Patient otherwise deemed at increased risk from this investigational rehabilitation program by their referring surgeon or physical therapist
* Patients who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in The Knee Injury and Osteoarthritis Outcome Score Pain Subscale | Baseline, Week 3
  Measured by the Pain Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Pain Subscale | Baseline, Month 6
  Measured by the Pain Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Pain Subscale | Baseline, Month 12
  Measured by the Pain Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Symptoms Subscale | Baseline, Week 3
  Measured by the Symptoms Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Symptoms Subscale | Baseline, Month 6
  Measured by the Symptoms Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Symptoms Subscale | Baseline, Month 12
  Measured by the Symptoms Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/sports and recreational activities Subscale | Baseline, Week 3
  Measured by the function/sports and recreational activities Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/sports and recreational activities Subscale | Baseline, Month 6
  Measured by the function/sports and recreational activities Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/sports and recreational activities Subscale | Baseline, Month 12
  Measured by the function/sports and recreational activities Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Quality of Life Subscale | Baseline, Week 3
  Measured by the Quality of life Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Quality of Life Subscale | Baseline, Month 6
  Measured by the Quality of life Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Quality of Life Subscale | Baseline, Month 12
  Measured by the Quality of life Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/daily living Subscale | Baseline, Week 3
  Measured by the function/daily living Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/daily living Subscale | Baseline, Month 6
  Measured by the function/daily living Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in The Knee Injury and Osteoarthritis Outcome Score Function/daily living Subscale | Baseline, , Month 12
  Measured by the function/daily living Knee injury and osteoarthritis score subscales (KOOS subscales). The KOOS survey is comprised of 42 questions. The questions are divided into 5 sub-categories: symptoms (7 questions), pain (9 questions), function/daily living (17 questions), function/sports and recreational activities (5 questions), and quality of life (4 questions). The total range for each sub-category is 0-100, making the total range for the whole survey 0-500. The higher the score, the worse the symptoms and pain/ higher difficulty in function.
Change in Visual Analogue Scale (VAS) Pain score | Baseline, Week 3
  VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Change in Visual Analogue Scale (VAS) Pain score | Baseline, Month 6
  VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Change in Visual Analogue Scale (VAS) Pain score | Baseline, Month 12
  VAS is a tool widely used to measure pain. A patient is asked to indicate his/her perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge (=VAS score). The total score range is 0 (no pain) to 10 (worst pain imaginable); the higher the score, the worse the pain.
Change in Active Range of Motion (AROM) | Baseline, Week 1
  AROM is measured using a goniometer (protractor that measures joint angles) to see how much the knee can bend and straighten on its own (without assistance). Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Active Range of Motion (AROM) | Baseline, Week 3
  AROM is measured using a goniometer (protractor that measures joint angles) to see how much the knee can bend and straighten on its own (without assistance). Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Active Range of Motion (AROM) | Baseline, Month 6
  AROM is measured using a goniometer (protractor that measures joint angles) to see how much the knee can bend and straighten on its own (without assistance). Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Active Range of Motion (AROM) | Baseline, Month 12
  AROM is measured using a goniometer (protractor that measures joint angles) to see how much the knee can bend and straighten on its own (without assistance). Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Passive Range of Motion (PROM) | Baseline, Week 1
  PROM is measured using a goniometer (protractor that measures joint angles) to see how far the knee can bend and straighten when moved by an external force. Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Passive Range of Motion (PROM) | Baseline, Week 4-6
  PROM is measured using a goniometer (protractor that measures joint angles) to see how far the knee can bend and straighten when moved by an external force. Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Passive Range of Motion (PROM) | Baseline, Month 6
  PROM is measured using a goniometer (protractor that measures joint angles) to see how far the knee can bend and straighten when moved by an external force. Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in Passive Range of Motion (PROM) | Baseline, Month 12
  PROM is measured using a goniometer (protractor that measures joint angles) to see how far the knee can bend and straighten when moved by an external force. Normal ROM at the knee is considered to be 0 degrees of extension (completely straight knee joint) to 135 degrees of flexion (fully bent knee joint).
Change in ACL-Return to Sport (ACL-RSI) Scale Score | Baseline, Week 3
  The ACL-RSI scale includes 12 questions on the patient's emotional well-being and confidence in his or her performance and risk appraisal. The scale, with scores ranging from 1 to 10, includes 5 questions on emotional well-being, 5 questions on confidence in physical performance, and 2 questions on the appraisal of risk. Higher scores indicate a more positive psychological response. The total score is determined by adding the values of the 12 responses and then calculating their relationship to 100 to obtain a percentage (0-100%).

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Gonzalez-Lomas, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request, Requests should be directed to Zachary.li@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.